CLINICAL TRIAL: NCT04375215
Title: Success of Selective Caries vs Stepwise Caries Removal Technique in Deep Carious Lesions- A Randomized Clinical Study
Brief Title: Selective Caries vs Stepwise Caries Removal Technique in Deep Carious Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VISHALPGIDS
Record Dates: First submitted 2020-04-24; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Caries

STUDY DESIGN:
Intervention Model Description: Prospective randomized clinical study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective caries removal to soft dentin (one step) (Active Comparator): In selective caries removal to soft dentine, after caries excavation application of liner will be done on pulpal floor. Teeth will then be filled with composite resin material.
  Interventions: Procedure: Selective caries removal
- Stepwise caries removal (two step) (Active Comparator): The stepwise caries removal is a two step procedure. The first step is similar to selective caries removal to soft dentin group. In the second step, after 6 months lesion will be re-entered to remove remaining carious tissue till firm dentin is encountered. Once all the caries is removed from floor of cavity a liner followed by final restoration with composite will be performed.
  Interventions: Procedure: Stepwise caries removal

INTERVENTIONS:
Procedure: Selective caries removal — After caries removal restoration of tooth will be performed
  Arms: Selective caries removal to soft dentin (one step)
Procedure: Stepwise caries removal — After caries removal restoration of tooth will be performed
  Arms: Stepwise caries removal (two step)

SUMMARY:
The aim of this clinical study is to compare and evaluate the Success of Selective Caries vs Stepwise Caries Removal Techniques in treatment of dental caries.

DETAILED DESCRIPTION:
The patient will be selected as per the pre-defined eligibility criteria. Written informed consent will be taken from each consenting participant. Initial caries excavation will be done under rubber dam isolation. The patient will then be randomly allocated to two groups: selective removal to soft dentin or stepwise caries removal. Composite restoration with glass ionomer liner will be then placed in both groups. Additional complete caries excavation will be done in the stepwise caries removal group after six months.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient in age range of 18yr-60yr
* Permanent mandibular posterior teeth with deep caries
* Caries extending to >3/4 of dentin with a layer of sound dentin between pulp and carious tissue as seen on radiograph
* Positive response to cold test and electric pulp test

Exclusion Criteria:

* Any general disease affecting the caries e.g. patient under head and neck radiotherapy
* Patients with immuno-compromised status
* Tooth with fracture line, cracks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Clinical success | Baseline to 12 months
  Clinical success will be judged by following criteria
  * Positive response on vitality test.
  * Absence of pain on percussion and any other signs and/or symptoms of irreversible pulpitis and pulp necrosis
  Criteria for failure will be
  * Negative response on pulp vitality test.
  * Tenderness to percussion and teeth exhibiting any clinical signs and/or symptoms of irreversible pulpitis and pulp necrosis.

SECONDARY OUTCOMES:
Radiographic Success | Baseline to 12 months
  Absence of periapical alterations (radiolucency at furcal or periapical region).

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Science, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No